CLINICAL TRIAL: NCT05899439
Title: Immune Function and the Progression to Type 1 Diabetes:
Brief Title: Immune Function and the Progression to T1D
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400709; PRO00043521 (Other: University of Florida); P01AI042288 (NIH)
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sample collections, mainly peripheral blood but also discarded clinical samples, will occur at clinics, research space, and special event spaces on the University of Florida campus and remotely via lab collection. Genetic analysis will be performed related to developing a genetic model for predicting type 1 diabetes in the general population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with diabetes age 0 to 100 years: People who have not been diagnosed with type 1 diabetes
  Interventions: Other: blood draw
- Subjects with type 1 diabetes age 0 to 100 years: People who have been diagnosed with type 1 diabetes
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — a peripheral blood draw

SUMMARY:
To elucidate the mechanisms by which type 1 diabetes-associated genes; IFIH1, TYK2, IKZF4, as well as total genetic risk, impart functional immunoregulatory abnormalities that result in expansion of self-reactive adaptive immune cells, defective regulatory/effector mechanisms in T cells, inflammatory antigen presenting cells, and abnormal immune function in T cells and B cells.

DETAILED DESCRIPTION:
Newly proposed studies will identify the inflammatory cues that draw immune cells into islets for disease initiation (Project 1); probe the motility of immune cells through inflamed vasculature to the target organ and antigen priming sites within secondary lymphatics (Project 2); and characterize the T1D-associated adaptive immune signatures in blood and immune tissues (Project 3).

The overall hypothesis of the renewed P01 states: 1) the impact of T1D-risk variants will vary by tissue, cell subset, and activation state, and 2) risk variants, cellular stress, and defects in immunologic pathways are key to engender the autoimmune destruction of pancreatic B-cells that results in T1D.

ELIGIBILITY:
Inclusion Criteria: able to have blood drawn -

Exclusion Criteria: none

-

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals age 0 to 100 with or without a diagnosis of type 1 diabetes and able/willing to have a blood draw
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2085-01-01 (Estimated); Study Completion 2085-01-01 (Estimated)

PRIMARY OUTCOMES:
the number of participants who become at risk for development of type 1 diabetes | through study completion, up to 25 years
  the number of participants who become at risk for development of type 1 diabetes
Genetic risk of type 1 diabetes | through study completion, up to 25 years
  the number of people in different genetic risk groups who develop type 1 diabetes

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kieran McGrail, Gainesville, Florida
  - The Ohio State University, Columbus, Ohio
  - Baylor College of Medicine, Center for Research Advancement - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
the data generated from the proposed studies will be presented at national or international conferences and published in a timely fashion. Investigators associated with this P01 have a record of publishing in pre-print servers and favoring open-access journals, when appropriate. The investigator will implement field standard, open-source tools including those developed by investigators on this proposal for data processing. Importantly, raw data, processed data, and metadata will be stored locally as well as deposited on public databases as detailed further below. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. Evidence of this is provided in the attached biosketches.